CLINICAL TRIAL: NCT03878472
Title: A Phase II Clinical Study of Neoadjuvant Therapy for Resectable Locally Advanced Gastric Cancer with PD-1 Antibody or in Combination with Apatinib ± S1±Oxaliplatin
Brief Title: Neoadjuvant Immunotherapy for Resectable Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIPASS2019
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; apatinib; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Neoadjuvant immunotherapy with PD-1 (Experimental)
  Interventions: Drug: SHR1210
- Neoadjuvant immunotherapy with PD-1+apatinib (Experimental)
  Interventions: Drug: SHR1210; Drug: Apatinib
- Neoadjuvant immunotherapy with PD-1+apatinib+S1 (Experimental)
  Interventions: Drug: SHR1210; Drug: Apatinib; Drug: S1
- Neoadjuvant immunotherapy with PD-1+apatinib+S1+Oxaliplatin (Experimental)
  Interventions: Drug: SHR1210; Drug: Apatinib; Drug: S1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: SHR1210 — The patients will receive at least two cycles of SHR-1210 (200 mg, invdrip d1) every two weeks and be accessed for operational suitability every two cycles.
Drug: Apatinib — The patients will received apatinib (250mg po qd) until 10 ± 2 days before surgery.
  Arms: Neoadjuvant immunotherapy with PD-1+apatinib; Neoadjuvant immunotherapy with PD-1+apatinib+S1; Neoadjuvant immunotherapy with PD-1+apatinib+S1+Oxaliplatin
Drug: S1 — The patients will received S1 (50 mg/m2, po, bid, d1-d10) every two weeks and be accessed for operational suitability every two cycles.
  Arms: Neoadjuvant immunotherapy with PD-1+apatinib+S1; Neoadjuvant immunotherapy with PD-1+apatinib+S1+Oxaliplatin
Drug: Oxaliplatin — The patients will receive at least two cycles of oxaliplatin (85 mg/m2 d1) every two weeks and be accessed for operational suitability every two cycles.
  Arms: Neoadjuvant immunotherapy with PD-1+apatinib+S1+Oxaliplatin

SUMMARY:
1. Target population: patients with resectable locally advanced gastric cancer (cT3-4bN+M0).
2. Primary objective:

(1) To evaluate the pathological remission rate (PRR) of PD-1 antibody monotherapy or in combination with anti-angiogenesis VEGFR2-TKI apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer.

(2) To evaluate the relationship between tumor pathological remission and biomarkers related to immunotherapy.

3. Secondary objectives:

1. To evaluate the imaging objective response rate (ORR), progression-free survival (PFS), and overall survival (OS) of PD-1 antibody alone or in combination with apatinib ± S1 ± Oxaliplatin in neoadjuvant therapy for locally advanced gastric cancer.
2. To evaluate the safety of PD-1 antibody or in combination with apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer.

Trial design: This is a monocenter, open, single arm, phase II study to evaluate the efficacy and safety of PD-1 antibody or in combination with apatinib ± S1 ± Oxaliplatin in neoadjuvant treatment of resectable locally advanced gastric cancer.

DETAILED DESCRIPTION:
Several important clinical trials including MAGIC, FLOT4, POET, RTOG 9904 and TOPGEAR have identified the efficacy and safety of neoadjuvant treatment in treating locally advanced GEJ cancer or gastric cancer.

patients with resectable locally advanced gastric cancer will receive neoadjuvant treatment of PD-1 antibody or in combination with apatinib ± S1 ± Oxaliplatin.

The investigators will shut down the study in advance, if situations below happens: 1) 1 treatment related death, >3 disease progression or >2 hyper-progressive disease happen during the first stage; 2) 2 treatment related death, >6 disease progression or >4 hyper-progressive disease happen during the whole study.

Patients with abnormal autoimmune status, unfavorable body function, factors impeding drug taking, absorption and metabolism will be excluded. Study participants with disease progression or severe/ intolerant toxicity during treatment will withdraw the study.

Hyper-progressive disease is defined as 1) progression 2) more than doubled growth rate 3) tumor volume increase >50% in 2 months after initialing the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years old, both genders, histologically documented gastric cancer.
2. Newly diagnosed locally advanced, potentially resectable disease without any prior antitumor treatment
3. clinically diagnosed stage T3-4bN+M0 according to ultrasound endoscopy or enhanced CT/MRI scan.
4. Eligible and reasonably suitable for potentially curative resection
5. Written (signed) informed consent.
6. Pathological tissue available
7. ECOG: 0-1.
8. Adequate organ function.
9. Willingness to provide blood and tissue samples for research purposes.
10. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
11. Female patients should not be pregnant or breast feeding.
12. Agree to take contraception measures during treatment and in 120 days after last dose of SHR-1210.
13. Life expectancy of at least 6 months.

Exclusion Criteria:

1. Patients with distant metastasis.
2. History of chemotherapy, radiation, immunotherapy, or radical resection of gastric cancer.
3. patients with active autoimmune disease or history of refractory autoimmune disease.
4. patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured locally tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ.
5. uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment.
6. patients who have digestive tract bleeding in 2 weeks before recruitment or with high risk of bleeding.
7. perforation / fistula of GI tract in 6 months before recruitment.
8. pulmonary disease history: interstitial pulmonary disease, non-infective pneumonitis, pulmonary fibrosis, acute pulmonary disease.
9. uncontrollable systemic diseases, including diabetes, hypertension etc.
10. severe chronic or active infections in need of systemic antibacterial, antifungal, or antiviral treatment, including TB or HIV, etc.
11. patients with untreated chronic hepatitis B or HBV DNA over 500 IU/ml or positive HCV RNA.
12. patients with any cardiovascular risk factors below: （1）cardiac chest pain occurring in 28 days before recruitment, defined as moderate pain that limits daily activity.

（2）pulmonary embolism with symptoms occurring in 28 days before recruitment. （3）acute myocardial infarction occurring in 6 months before recruitment. （4）any history of heart failure reaching grade 3/4 of NYHA in 6 months before recruitment.

（5）ventricular arrhythmias of Grade 2 or grater in 6 months before recruitment, or accompanied by supraventricular tachyarrhythmias requiring medical treatment.

（6）cerebrovascular accident within 6 months before recruitment. 14. patients with peripheral neuropathy NCI CTC AE grade 1, except those with only deep tendon reflex disappearing.

15. moderate or severe renal injury [creatinine clearance rate≤50 ml/min (according to Cockcroft & Gault equation)], or Scr>ULN.

16. dipyrimidine dehydrogenase (DPD) deficiency. 17. allergic to any drug in this study. 18. history of allogeneic stem cell transplantation or organ transplantation. 19. use of steroids (dosage>10mg/d prednisone) or other systemic immune suppressive therapy in 14 days before recruitment, except patients treated with regimens below: a. steroids for hormone replacement (dosage>10mg/d prednisone); b. steroids for local application with little systemic absorption; c. short -term (≤ 7 days) steroids for preventing allergy or vomiting.

20. vaccinated with live vaccine in 4 weeks before recruitment. 21. for patients with uncontrolled epilepsy, CNS diseases or history of mental disorder, researchers should evaluate whether their diseases will impede their signing of informed consent or compliance of treatment.

22. existing of potential situation which will impede drug administration or affect toxicity analysis or alcohol/ drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Pathological remission rate (PRR) rate of PD-1 antibody monotherapy or in combination with anti-angiogenesis VEGFR2-TKI apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer. | 5 months after the last subject participating in
  The pathological response was calculated according to the proportion of residual viable tumor cells in the tumor bed. Complete pathological response (CPR) was defined as no residue tumor cells. Major pathological response (MPR) was defined as less than 10% residue tumor cells.
Immunotherapy-related biomarkers | 5 months after the last subject participating in
  To evaluate the relationship between tumor pathological remission and immunotherapy related biomarkers, including tumor genome, tumor microenvironment and host immune system response biomarkers.

SECONDARY OUTCOMES:
objective response rate (ORR) of PD-1 antibody monotherapy or in combination with anti-angiogenesis VEGFR2-TKI apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer. | Time Frame: 36 months after the last subject participating in
  rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1. However, responses do not require confirmation according to RECIST v 1.1. ORR was evaluated by chest, abdominal & pelvic CT/MRI.
progression free survival (PFS)of PD-1 antibody monotherapy or in combination with anti-angiogenesis VEGFR2-TKI apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer. | Time Frame: 36 months after the last subject participating in
  PFS is defined as time interval from recruitment to tumor progression. Tumor progression is defined as below: 1) tumor re-occurrence, 2) death, 3) censoring, and 4) beginning to use any other anti-tumor medicines.
overall survival (OS) of PD-1 antibody monotherapy or in combination with anti-angiogenesis VEGFR2-TKI apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer. | Time Frame: 36 months after the last subject participating in
  OS is defined as time interval from recruitment to all-caused death or censoring.
safety as measured by the rate of adverse events (AEs), laboratory abnormalities, dose adjustment, discontinuation of administration, early discontinuation of the study drug, and delay to surgery. | Time Frame: 1 month after the last date of treatment
  Adverse events (AEs) of neoadjuvant therapy will be graded and documented according to NCI-CTCAE v4.0 from the beginning of treatment to 1 months after the last date of treatment. Documentary will include severity, lasting period and occurrence time. Main AEs include vomiting, diarrhea, anemia, leukopenia, thrombocytopenia, hand-foot syndrome, epidermal capillary hyperplasia, immune related adverse events (including pneumonia, interstitial lung disease, AST/ALT elevations, rash, diarrhea, hypothyroidism and hyperthyroidism) and hyper-progressive tumor.
  AEs of surgery refer to complications which happen during or in 30 days after operation. Severe complications after operation such as abdominal or GI tract bleeding, anastomotic fistula, pancreatic fistula of grade B or above, incision complications (infection, bleeding, rupture) will be observed and classified by Clavien-Dindo grading.
R0 resection rate | 5 months after the last subject participating in
  To evaluate the R0 resection rate of PD-1 antibody monotherapy or in combination with anti-angiogenesis VEGFR2-TKI apatinib ± S1 ± Oxaliplatin in neoadjuvant (preoperative) treatment of resectable locally advanced gastric cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong univertisy, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided